CLINICAL TRIAL: NCT05444543
Title: Effectiveness of Cycling of Topical Steroid Therapy in Maintaining Clinical and Histologic Remission in Eosinophilic Esophagitis
Brief Title: Cycling of Topical Steroids for Treatment of EoE (Eosinopilic Esophagitis)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Thomas J Sferra, MD, Chief of Pediatric Gastroenterology Hepatology and Nutrition, University Hospitals Cleveland Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20210671
Record Dates: First submitted 2022-06-28; First posted 2022-07-06 (Actual); Results first posted 2024-11-07 (Actual); Last update posted 2024-11-07 (Actual); Status verified 2024-10

CONDITIONS: Eosinophilic Esophagitis
Keywords: Fluticasone; Budesonide; Adolescent; Cycling
MeSH Terms: conditions — Eosinophilic Esophagitis | interventions — Fluticasone; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention): Participants in this arm will continue with their normal standard of care regimen of daily topical steroids
- Intervention (Experimental): Participants in this arm will cycle their topical steroid therapy in a three-months on three-months off fashion
  Interventions: Drug: Fluticasone Propionate; Drug: Budesonide

INTERVENTIONS:
Drug: Fluticasone Propionate — Participants will cycle topical steroid in a three-months on three-months off fashion
  Arms: Intervention
Drug: Budesonide — Participants will cycle topical steroid in a three-months on three-months off fashion
  Arms: Intervention

SUMMARY:
The purpose of our research study is to assess whether patients with EoE who have achieved control of their disease on topical Fluticasone or Budesonide are able to cycle or take breaks from their treatment with continued remission of their EoE. There will be 30 participants enrolled in this study. There will be 15 patients who will stay on steroid therapy every day and 15 patients who will cycle their steroid therapy on and off to help us compare the two groups. The cycling group will cycle their steroid therapy in a three-months on three-months off fashion.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients between 4-18 years of age with EoE followed by the Division of Pediatric Gastroenterology, Hepatology and Nutrition at Rainbow Babies and Children's Hospital
* Patients who are currently on treatment with topical corticosteroids and scheduled for an upcoming endoscopy as part of their routine clinical care (to be used as EGD1) within 3 months of enrollment date
* Patients who have achieved documented clinical and endoscopic remission using topical steroids as evidenced by EGD

Exclusion Criteria:

* Patients who are not responsive to topical corticosteroid treatment for their EoE as evidenced by failure to obtain clinical or endoscopic remission on any pervious screening EGD
* Patients less than 4 years of age and older than 18 years of age at the time of recruitment
* Patients with history of or current diagnosis of esophageal strictures

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 23 (Actual)
Dates: Start 2021-11-17 (Actual); Primary Completion 2023-10-13 (Actual); Study Completion 2023-10-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Sferra, MD, Principal Investigator — University Hospitals Cleveland Medical Center; Nuphar Lendner, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Intervention
Started | 11 | 12
Completed | 9 | 10
Not Completed | 2 | 2
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Failed to achieve initial remission on therapy | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Family relocating at a distance from study site | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Intervention | Total
Number analyzed (Participants) | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: Years] | 11.6 (3.4) | 15.5 (3.2) | 12.5 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 5 | 9
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 11 | 11 | 22
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 11 | 10 | 21
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 2 | 2

OUTCOME MEASURES:

1. Primary Outcome: Percent of Patients in Remission at One Year as Measured by EGD
Description: The outcome measure is the number of participants who maintained remission (less than or equal to 15 eosinophils per high powered field in esophageal biopsies) for one year after demonstration of a therapeutic effect of topical steroid therapy.
Time Frame: up to one year
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 9 | 10
Participants | 5 | 1
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p = 0.57, Chi-squared; Odds Ratio (OR) = 0.089

2. Secondary Outcome: Number of Patients Who Report Adverse Events as Measured by Patient Report
Time Frame: up to 12 months
Population: Includes all enrolled participants, number of participants reporting an adverse event
Measure: Count of Participants; unit: Participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 11 | 12
Participants | 1 | 1
Statistical Analysis 1: Comparison: Control vs Intervention; Test type: Superiority; p > 0.99, Chi-squared; Odds Ratio (OR) = 1.1

3. Secondary Outcome: Number of Patients Who Develop Subclinical Adrenal Insufficiency as Measured by Blood Work
Description: Subclinical adrenal insufficiency was defined as a morning cortisol level less than 10.0 micrograms per deciliter. One low level at anytime during the study period was recorded as an insufficient level.
Time Frame: up to 12 months
Population: Includes all enrolled participants and those who had cortisol levels obtained at the scheduled time.
Measure: Number; unit: participants
Arm/Group | Control | Intervention
Number analyzed (Participants) | 7 | 12
participants | 4 | 6

4. Other Pre Specified Outcome: Change in Quality of Life as Measured by Modified-PedsQL™ Eosinophilic Esophagitis Module Child Self-Report Item Content
Description: 14 item questionnaire where patients either agree or disagree
Time Frame: Baseline, 3 months, 6 months, 12 months
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Percent of Patients With Elevated IL-13 as Measured by Biopsy
Time Frame: up to 12 months
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Percent of Patients With Elevated Eotaxin as Measured by Biopsy
Time Frame: up to 12 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Control | Intervention
All-Cause Mortality (participants affected / at risk) | 0/11 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/11 | 0/12
Other Adverse Events (participants affected / at risk) | 2/11 | 2/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=11) | Intervention (N=12)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1)
Candidiasis of mouth (Infections and infestations) | 1 (1) | 0 (0)
Ulcer of mouth (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-12): https://cdn.clinicaltrials.gov/large-docs/43/NCT05444543/Prot_SAP_000.pdf